CLINICAL TRIAL: NCT04239742
Title: F18-PSMA-1007 PET for Early Biochemical Recurrence of Prostate Cancer, Comparison With 18F-Fluciclovine
Brief Title: F18-PSMA-1007 PET for Early Biochemical Recurrence of Prostate Cancer
Acronym: PROPER-ABX
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Radboud University Medical Center (Other)
Collaborators: ABX advanced biochemical compounds GmbH (Industry); Radboud Translational Medicine (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NL65593.091.18
Record Dates: First submitted 2020-01-13; First posted 2020-01-27 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Prostate Cancer Recurrent
Keywords: 18F-PSMA-1007; 18F-Fluciclovine

STUDY DESIGN:
Intervention Model Description: every individual gets two diagnostic PET CT scans within 2 weeks apart.
Masking Description: scans will be anonymized for study outcome assessment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- 18F-PSMA PET/CT and 18F-Fluciclovin PET/CT (Experimental): patients undergo an 18F-PSMA PET/CT scan and an 18F-Fluciclovin PET/CT scan, within a time frame of two weeks.
  Interventions: Diagnostic Test: F18-fluciclovine PET/CT; Diagnostic Test: F18-PSMA-1007 PET/CT

INTERVENTIONS:
Diagnostic Test: F18-fluciclovine PET/CT — 370 MBq ±10% 18F-Fluciclovin + low-dose CT scan, from skull base to pelvis.
  Other Names: Axumin scan
Diagnostic Test: F18-PSMA-1007 PET/CT — 4 MBq/kg ±10% F18-PSMA + low-dose CT scan, from skull base to pelvis
  Other Names: PSMA scan

SUMMARY:
18F-PSMA-1007 is a new radiopharmaceutical for the detection of prostate cancer with potential benefits over the registered 18F-Fluciclovine (Axumin). The main potential benefit is the higher detection rate of PSMA compared to Fluciclovin in the low PSA range. It may therefore be more sensitive in detecting local disease in case of biochemical recurrens. The investigators aim to compare the detection efficacy of 18F-PSMA-1007 to 18F-Fluciclovin in prostate cancer patients with biochemical recurrence (PSA levels 0.2-5 ng/ml).

DETAILED DESCRIPTION:
Rationale: 18F-PSMA-1007 is a new radiopharmaceutical for detection of prostate cancer with potential benefits over 18F-Fluciclovine, such as higher detection rates at low PSA levels and small lesions, lower bone marrow uptake and higher tumour-background ratio. Therefore, 18F-PSMA-1007 PET may be more sensitive in detecting local recurrence and metastases of prostate cancer. However, Fluciclovine is a registered tracer, whereas PSMA-1007 is not registered, and therefore there is pressure to use fluciclovine instead of PSMA-1007. Therefore more comparative data are urgently needed.

Objective: Main objective is to compare detection efficacy of 18F-PSMA-1007 PET-CT to 18F-Fluciclovine, in patients with early biochemical recurrence of prostate cancer.

Study design: Comparative phase II diagnostic study Study population: 50 males >18 years, with biochemical recurrence of prostate cancer and PSA-levels between 0.2-5.0 ng/mL. About 25 of the patients must have PSA-levels between 0.2-1.0 ng/mL. Contra-indications: claustrophobia, inability to lay still for the duration of the exam. Already established local recurrence in the prostate is not a contra-indication for study participation.

Intervention: 50 patients who already were referred by their treating physician for PET/CT will receive both an 18F-PSMA-1007 PET-CT (90 minutes post injection) and an 18F-Fluciclovine PET-CT (<15 minutes post injection). Injected dose of the 18F-PSMA-1007 will be 4 MBq/kg ±10%. The injected dose of 18F-Fluciclovine is 370 MBq ±10%.

Analysis: A clinical report is made of both the 18F-PSMA-1007 PET-CT scan and 18F-Fluciclovine PET-CT scan. For further analysis in the study all data will be anonymized, and will be blindly scored by two nuclear medicine physicians. The number of PET-positive lesions (judged to be prostate cancer, of course PET positive lesions referring to different processes like inflammation will not be taken intob account, this is oart of the PET-reading process) per area are separately scored for both tracers. Lesions will be scored on a 5-point scale ranging from most probably benign to most probably malignant. Follow-up data of the patients, to determine the eventual outcome, will be extracted from their medical file. An expert panel will eventually decide which lesions are considered to be metastases using all available follow-up data.

ELIGIBILITY:
Inclusion Criteria:

* Males ≥ 18 years
* Histologically proven adenocarcinoma of the prostate
* Prior local treatment with curative intent
* Biochemical recurrence with (rising) PSA-levels of 0.2-5.0 ug/L
* Referred by urologist for PET/CT for localization of the recurrence
* PSA level determined <8 weeks before study participation
* Willing to sign informed consent

Exclusion Criteria:

* Contra-indications for PET-CT: claustrophobia or inability to lay still for the duration of the exam.
* Other cancer <2 years prior to biochemical recurrence of prostate cancer

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-01-02 (Actual); Primary Completion 2022-01 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
Detection efficacy of the two PET-tracers on a per patient level | Follow-up duration is 6 months.
  Comparisson of number of patients with a positive scan
Detection efficacy of the two PET-tracers on a per lesion level | Follow-up duration is 6 months.
  Comparisson of number of positive lesions

SECONDARY OUTCOMES:
Quantitative analysis | 6 months
  tumour background ratio, SUV (of tumor and normal organs)
Comparing specificity | 6 months
  where the reference is consensus by the expert panel using all available information including 6 months follow up data (PSA-values; absolute and doublind time, pathology reports of suspected prostate cancer lesions, prostate-cancer targeted imaging by PET CT, MRI, CT or bone scan).
Sensitivity per area, local recurrence | 6 months
  local recurrence, where the reference test is consensus by the expert panel using 6 months available clinical follow-up data.
Sensitivity per area, locoregional lymph nodes | 6 months
  locoregional lymph nodes, where the reference test is consensus by the expert panel using 6 months available clinical follow-up data.
Sensitivity per area, distant lymph nodes | 6 months
  Distant lymph nodes, where the reference test is consensus by the expert panel using 6 months available clinical follow-up data.
Sensitivity per area, bone metastases | 6 months
  Bone metastases, where the reference test is consensus by the expert panel using 6 months available clinical follow-up data.
Sensitivity per area, extraskeletal organ metastases, where the reference test is consensus by the expert panel using 6 months available clinical follow-up data. | 6 months
  Extraskeletal organ metastases

CONTACTS AND LOCATIONS:
Overall Officials: James Nagarajah, MD, PhD, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboudumc, Nijmegen, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Loeff CC, van Gemert W, Prive BM, van Oort IM, Hermsen R, Somford DM, Nagarajah J, Heijmen L, Janssen MJR. [18F]PSMA-1007 PET for biochemical recurrence of prostate cancer, a comparison with [18F]Fluciclovine. EJNMMI Rep. 2024 Nov 27;8(1):38. doi: 10.1186/s41824-024-00228-2. PMID 39592501